CLINICAL TRIAL: NCT00609466
Title: A Randomized, Double-blind, Parallel-group, Multi-center, Active- and Placebo-controlled Trial to Evaluate the Analgesic Efficacy and Safety of Multiple Doses of CG5503 IR for Postoperative Pain Following Bunionectomy
Brief Title: A Trial to Evaluate CG5503 Efficacy and Safety in Acute Pain After Bunionectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 574139
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Results first posted 2009-11-25 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Bunionectomy; Pain; Postoperative Pain; Acute Pain
Keywords: Opioid; Central acting analgesic; CG5503 IR; Postoperative pain; Bunionectomy; Morphine; Placebo
MeSH Terms: conditions — Pain; Pain, Postoperative; Acute Pain | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): CG5503 IR 75mg 4 to 6 hourly for 72 hours
  Interventions: Drug: CG5503 IR
- 2 (Active Comparator): Morphine IR 30 mg 4 to 6 hourly for 72 hours
  Interventions: Drug: Morphine
- 3 (Placebo Comparator): Matching placebo 4 to 6 hourly for 72 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CG5503 IR — 75mg IR 4 - 6 hourly Total: 72 hours
  Arms: 1
Drug: Morphine — Morphine 30 mg IR 4 - 6 hourly Total: 72 hours
  Arms: 2
Drug: Placebo — Placebo; 4 - 6 hourly; Total: 72 hours
  Arms: 3

SUMMARY:
The main objective of this trial is to demonstrate the efficacy and safety of multiple-dose application of oral application of CG5503 IR 75mg compared to placebo and to assess safety and tolerability of CG5503 IR 75mg in subjects following bunionectomy.

This trial was performed based on a previously performed double-blind, placebo-controlled, multiple-dose trial in the same indication investigating 3 dose strengths CG5503 IR (50, 75 and 100 mg) published under PMID: 18851776.

DETAILED DESCRIPTION:
Subjects undergoing bunionectomy often experience moderate to severe acute pain post-surgery. Normally such pain is controlled when subjects receive repeated doses of opioid analgesics. However, opioid therapy is commonly associated with side effects such as nausea, vomiting, sedation, constipation, addiction, tolerance, and respiratory depression. CG5503, a newly synthesized drug with an immediate release (IR) formulation, also acts as a centrally acting pain reliever but has a dual mode of action. The aim of this trial is to investigate the effectiveness (level of pain control) and safety (side effects) of CG5503 IR 75mg compared with no drug (placebo) or one dose of morphine (an opioid commonly used to treat post-surgical pain). This trial is a randomized, double-blind (neither investigator nor patient will know which treatment was received), active- and placebo-controlled, parallel-group, multicenter trial to evaluate the treatment of acute pain after bunionectomy. The trial will include a blinded 72 hour inpatient phase immediately following bunionectomy, during which subjects will be treated with either 75-mg CG5503 IR, a placebo, or 30-mg morphine, and pain relief will be periodically assessed. Assessments of pain relief include the pain intensity numeric rating scale (PI), pain relief numeric rating scale (PAR), and patient global impression of change scale (PGIC). Safety evaluations include monitoring of adverse events, physical examinations, and clinical laboratory tests. Venous blood samples will be collected for the determination of serum concentrations of CG5503 and morphine. The alternative trial hypothesis is that at least 1 dose strength of CG5503 will be different from placebo in controlling pain at 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 18 and 80 years of age;
* Scheduled to undergo primary unilateral first metatarsal bunionectomy;
* Anesthesiological and surgical procedures performed according to protocol;
* Moderate or severe baseline pain following bunionectomy on a VRS within 9 hours of termination of the continuous popliteal sciatic block or systemic analgesia;
* Pain following bunionectomy of at least 4 on an 11-point NRS within 9 hours of termination of the continuous popliteal sciatic block or systemic analgesia; American Society of Anesthesiologists (ASA) classification I-III.

Exclusion Criteria:

* History of seizure disorder;
* History of alcohol, medication or drug dependency, unstable psychological personality requiring intermittent or permanent treatment; severely impaired renal function, moderately or severely impaired hepatic function;
* Contraindications to, or history of allergy or hypersensitivity to CG5503, oxycodone, morphine, fentanyl hydrocodone, acetaminophen, heparin, or any compound planned to be used during the anesthesia, or their excipients;
* Pre-operative use within 12h prior to surgery or peri-operative use of non- steroidal anti-inflammatory drugs (NSAIDs);
* Treated regularly with opioid analgesic or NSAIDs within 30 days prior to screening;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2007-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E Daniels, DO, Principal Investigator — Premier Research Group (formerly SCIREX Corporation)
Locations (6):
- United States (6):
  - Site 104, Pasadena, Maryland
  - Site 101, Austin, Texas
  - Site 102, Houston, Texas
  - Site 105, San Antonio, Texas
  - Site 103, San Marcos, Texas
  - Site 106, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for this in-patient, multicenter study occurred between 04 September 2007 and 11 December 2007.
Pre-assignment Details: The trial consisted of a Screening Period (Day -28 up to the first surgical incision on Day -1), a Surgical Period (Day -1 to Day 1 at approximately 03:00 h.), a Qualification Period (Day 1), a Double-Blind Treatment Period (Day 1 up to Day 4), and a Follow-up Period (Day 8 up to Day 18).
Groups:
- CG5503: CG5503 IR 75mg 4-6 hourly
- Morphine: Morphine IR 30mg 4 to 6 hourly
- Placebo: Matching Placebo 4 to 6 hourly
Period: Overall Study
Arm/Group | CG5503 | Morphine | Placebo
Started | 96 | 96 | 99
Completed | 94 | 90 | 95
Not Completed | 2 | 6 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Adverse Event | 2 | 3 | 1
Not completed — Lack of Efficacy | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CG5503 | Morphine | Placebo | Total
Number analyzed (Participants) | 96 | 96 | 99 | 291
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1 | 2
  Between 18 and 65 years | 94 | 88 | 90 | 272
  >=65 years | 2 | 7 | 8 | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 44.6 (12.58) | 43.7 (14.19) | 43.8 (13.93) | 44.0 (13.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 73 | 88 | 244
  Male | 13 | 23 | 11 | 47
Region of Enrollment [Number; unit: participants]
  United States | 96 | 96 | 99 | 291

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Differences Relative to the Baseline Pain Intensity.
Description: Pain Intensity assessed at predefined time points over a 48 hour period using an 11-point Numeric Rating Scale (NRS) where a score of zero indicates "no pain" and a score of ten indicates "pain as bad as you can imagine". Differences calculated as [baseline-post baseline] at each predefined time point. The theoretical maximum range of Sum of pain intensity differences (SPID48) is from -480 (indicative of an increase in pain) to 480 (indicative of a decrease in pain).
Time Frame: Baseline value to 48 hours after first study drug intake.
Population: Intention to Treat - randomized subjects who were dosed and had a baseline pain intensity assessment. Last observation carried forward was used.
Measure: Mean (Standard Deviation); unit: units
Arm/Group | CG5503 | Morphine | Placebo
Number analyzed (Participants) | 96 | 93 | 96
units | 46.2 (130.83) | 102.5 (153.26) | -17.5 (111.27)
Statistical Analysis 1: Comparison: CG5503 vs Placebo; Null hypothesis of no treatment difference; Test type: Superiority or Other; p < 0.0001, ANCOVA — No multiplicity adjustment used; ANCOVA with treatment and centre as fixed effects and baseline pain as covariate; Least square mean = 70.8, 95% CI [35.9 to 105.6]

2. Secondary Outcome: Number of Participants Using Rescue Medication
Description: Number of participants who used at least one dose of rescue medication during the 72 hour double blind period.
Time Frame: Baseline up to 72 hours after first study drug intake
Population: Intention to treat (ITT) and Last Observation Carried Forward (LOCF)
Measure: Number; unit: participants
Arm/Group | CG5503 | Morphine | Placebo
Number analyzed (Participants) | 96 | 93 | 96
participants | 62 | 46 | 82
Statistical Analysis 1: Comparison: CG5503 vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank — Test for time (in hours) to first rescue medication use. No multiplicity adjustment; Adjusted for site

3. Secondary Outcome: Total Pain Relief (TOTPAR)
Description: Total pain relief (TOTPAR) in the 48 hour period from the first dose of study drug. The subject was to indicate pain relief at rest in response to the following question: How much relief have you had from your starting pain? None = 0, A little = 1, Some = 2, A lot = 3 and Complete = 4. The theoretical maximum range of Total pain relief (TOTPAR)48 is from 0 (indicative of no pain relief) to 192. The higher the value the better the pain relief.
Time Frame: Baseline to 48 hours after first study drug intake
Population: Intention to treat(ITT)and Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: units
Arm/Group | CG5503 | Morphine | Placebo
Number analyzed (Participants) | 96 | 93 | 96
units | 79.2 (49.63) | 81.6 (56.30) | 41.8 (50.88)
Statistical Analysis 1: Comparison: CG5503 vs Placebo; Null hypothesis of no treatment difference; Test type: Superiority or Other; p < 0.0001, ANCOVA — No multiplicity adjustment used; ANCOVA with treatment and centre as fixed effects and baseline pain as covariate; Least square mean = 37.5, 95% CI [22.7 to 52.2]

4. Secondary Outcome: Sum of Pain Intensity Differences Over 6 Hours (SPID6) Relative to the Baseline Pain Intensity
Description: Pain Intensity assessed at predefined time points over a 6 hour period using an 11-point Numeric Rating Scale (NRS) where a score of zero indicates "no pain" and a score of ten indicates "pain as bad as you can imagine". Differences calculated as [baseline-post baseline] at each predefined time point. The theoretical maximum range of Sum of pain intensity differences (SPID6) is from -60 (indicative of an increase in pain) to 60 (indicative of a decrease in pain).
Time Frame: Baseline to 6 hours after intake of first study drug
Population: Intention to treat(ITT) and Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: units
Arm/Group | CG5503 | Morphine | Placebo
Number analyzed (Participants) | 96 | 93 | 96
units | 8.0 (13.51) | 8.0 (15.59) | -1.2 (13.10)
Statistical Analysis 1: Comparison: CG5503 vs Placebo; Null hypothesis of no treatment difference; Test type: Superiority or Other; p < 0.0001, ANCOVA — No multiplicity adjustment used; ANCOVA with treatment and centre as fixed effects and baseline pain as covariate; Least square means = 9.9, 95% CI [6.2 to 13.6]

5. Secondary Outcome: Sum of Pain Intensity Differences Over 12 Hours (SPID12) Relative to the Baseline Pain Intensity
Description: Pain Intensity assessed at predefined time points over a 12 hour period using an 11-point Numeric Rating Scale (NRS) where a score of zero indicates "no pain" and a score of ten indicates "pain as bad as you can imagine". Differences calculated as [baseline-post baseline] at each predefined time point. The theoretical maximum range of Sum of pain intensity differences (SPID12) is from -120 (indicative of an increase in pain) to 120 (indicative of a decrease in pain).
Time Frame: Baseline to 12 hours after first study drug intake
Population: Intention to treat (ITT) and Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: units
Arm/Group | CG5503 | Morphine | Placebo
Number analyzed (Participants) | 96 | 93 | 96
units | 14.4 (28.89) | 17.9 (32.12) | -4.7 (24.82)
Statistical Analysis 1: Comparison: CG5503 vs Placebo; Null hypothesis of no treatment difference; Test type: Superiority or Other; p < 0.0001, ANCOVA — No multiplicity adjustment used; ANCOVA with treatment and centre as fixed effects and baseline pain as covariate; Least square mean = 20.6, 95% CI [13.2 to 28.0]

6. Secondary Outcome: Sum of Pain Intensity Differences Over 24 Hours (SPID24) Relative to the Baseline Pain Intensity
Description: Pain Intensity assessed at predefined time points over a 24 hour period using an 11-point Numeric Rating Scale (NRS) where a score of zero indicates "no pain" and a score of ten indicates "pain as bad as you can imagine". Differences calculated as [baseline-post baseline] at each predefined time point. The theoretical maximum range of Sum of pain intensity differences (SPID24) is from -240 (indicative of an increase in pain) to 240 (indicative of a decrease in pain).
Time Frame: Baseline to 24 hours after first study drug intake
Population: Intention to treat (ITT)and Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: units
Arm/Group | CG5503 | Morphine | Placebo
Number analyzed (Participants) | 96 | 93 | 96
units | 22.3 (60.17) | 41.3 (68.96) | -10.7 (51.28)
Statistical Analysis 1: Comparison: CG5503 vs Placebo; Null hypothesis of no treatment difference; Test type: Superiority or Other; p < 0.0001, ANCOVA — No multiplicity adjustment used; ANCOVA with treatment and centre as fixed effects and baseline pain as covariate; Least square mean = 36.4, 95% CI [20.7 to 52.0]

7. Secondary Outcome: Sum of Pain Intensity Differences Over 72 Hours (SPID72) Relative to the Baseline Pain Intensity
Description: Pain Intensity assessed at predefined time points over a 72 hour period using an 11-point Numeric Rating Scale (NRS) where a score of zero indicates "no pain" and a score of ten indicates "pain as bad as you can imagine". Differences calculated as [baseline-post baseline] at each predefined time point. The theoretical maximum range of Sum of pain intensity differences (SPID72) is from -720 (indicative of an increase in pain) to 720 (indicative of a decrease in pain).
Time Frame: Baseline to 72 hours after first intake of study drug
Population: Intention to treat (ITT) and Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: units
Arm/Group | CG5503 | Morphine | Placebo
Number analyzed (Participants) | 96 | 93 | 96
units | 78.4 (212.05) | 174.1 (242) | -19.1 (179.48)
Statistical Analysis 1: Comparison: CG5503 vs Placebo; Null hypothesis of no treatment difference; Test type: Superiority or Other; p = 0.0002, ANCOVA — No multiplicity adjustment used; ANCOVA with treatment and centre as fixed effects and baseline pain as covariate; Least square means = 108.2, 95% CI [51.9 to 164.5]

ADVERSE EVENTS:
Arm/Group | CG5503 | Morphine | Placebo
Serious Adverse Events (participants affected / at risk) | 0 | 1 | 0
Other Adverse Events (participants affected / at risk) | 69 | 85 | 47
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | CG5503 | Morphine | Placebo
Stevens Johnson Syndrome (Skin and subcutaneous tissue disorders) | 0/96 (0) | 1/96 (1) | 0/99 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | CG5503 | Morphine | Placebo
Nausea (Gastrointestinal disorders) | 46/96 (79) | 65/96 (147) | 24/99 (34)
Vomiting (Gastrointestinal disorders) | 21/96 (40) | 56/96 (156) | 4/99 (8)
Constipation (Gastrointestinal disorders) | 11/96 (11) | 13/96 (13) | 5/99 (6)
Dry Mouth (Gastrointestinal disorders) | 6/96 (8) | 8/96 (8) | 0/99 (0)
Dizziness (Nervous system disorders) | 29/96 (62) | 23/96 (39) | 17/99 (25)
Headache (Nervous system disorders) | 19/96 (27) | 28/96 (38) | 24/99 (32)
Somnolence (Nervous system disorders) | 12/96 (17) | 13/96 (15) | 4/99 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 15/96 (29) | 20/96 (25) | 0/99 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 4/96 (5) | 17/96 (21) | 2/99 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1/96 (1) | 7/96 (7) | 2/99 (2)
Alanine aminotransferase increased (Investigations) | 1/96 (1) | 7/96 (7) | 2/99 (2)
Aspartate aminotransferase increased (Investigations) | 1/96 (1) | 5/96 (5) | 1/99 (1)
Gamma glutamyl transferase increased (Investigations) | 1/96 (1) | 7/96 (7) | 4/99 (4)
Decreased appetite (Metabolism and nutrition disorders) | 0/96 (0) | 6/96 (6) | 0/99 (0)

LIMITATIONS AND CAVEATS:
Lortab (hydrocodone/acetaminophen) was allowed as rescue medication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Grünenthal GmbH reserves the right to review any publication pertaining to the trial before it is submitted for publication. Neither Grünenthal nor the investigator has the right to prohibit publication unless publication can be shown to affect possible patent rights.